CLINICAL TRIAL: NCT02139917
Title: Effects of a Transitional Palliative Care Model on Patients With ESRF
Brief Title: Effects of a Transitional Palliative Care Model on Patients With End-stage Renal Failure
Acronym: ESRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, TAM Mee Ling Bonnie, Clinical Associate, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23 January 2014
Record Dates: First submitted 2014-05-05; First posted 2014-05-16 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Palliative Care; Renal Failure, End-stage
Keywords: transitional palliative care; end stage renal failure
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transitional Palliative Care (Experimental): Transitional palliative care include:-
  * telephone follow up for early identification of signs and symptoms
  * home visit for spiritual support
  Interventions: Behavioral: Transitional community based palliative care
- Customary care (No Intervention): Customary care receive care :-
  * hospital based medical follow up
  * general nursing assessment and advice

INTERVENTIONS:
Behavioral: Transitional community based palliative care — transitional palliative care include:-
  * telephone follow up for early identification of signs and symptoms
  * relief of signs and symptoms encountered
  * home visit with spiritual support
  Other Names: Transitional palliative care
  Arms: Transitional Palliative Care

SUMMARY:
Primary aim:

1. To compare the effects of customary care and an interventional Home-based Palliative Renal Program (HBPRP) for ESRF patients
2. To compare the effects of customary care and Home-based Palliative Program (HBPP) for ESRF patients

   Secondary aim:
3. To explore the lived experiences of patients with ESRF. Hypothesis The transitional renal palliative care model is associated with decreased in unscheduled hospital readmission, reduce length of stay as well as improved quality of life for patients with end-stage renal failure.

DETAILED DESCRIPTION:
Objectives

Related to the primary aim:

1. Are there differences in healthcare utilization between the ESRF patients in the customary care group and those in the HBPRP group; in the HBPRP group and HBPP group?
2. Are there differences in evaluated health outcomes (functional status, symptom intensity, and satisfaction with care) between the customary care group and the HBPRP group ; in the HBPRP group and HBPP group?
3. Are there differences in perceived health outcomes (quality of life, caregiver burden) between the customary care group and the HBPRP group; in the HBPRP group and HBPP group?

   Related to the secondary aim:
4. How are the lived experiences compared and contrasted between the customary care group and the HBPRP group; in the HBPRP group and HBPP group?

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic kidney disease and diabetic mellitus with Creatinine ≥350 milli mole (uM) or those without diabetic mellitus with Creatinine ≥450 milli mole (uM) who refused renal replacement therapy (RRT);
* Patient not suitable for long term renal replacement therapy (RRT) after assessment by renal team (e.g. multiple co morbidities, poor functional status and social support)
* Identified as ESRF patient eligible for palliative care without prior renal replacement therapy
* Ability to speak Cantonese
* Living within the hospital service area
* Ability to be contacted by phone

Exclusion Criteria:

* Discharged to nursing home or other institution
* Inability to communicate
* Cognitive impairment, mini mental stage examination (MMSE) < 20
* Diagnosed with severe psychiatric disorders such as schizophrenia and bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-08; Primary Completion 2017-09 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Healthcare utilization composite - The dates of re-hospitalizations, length of stay, and number of other hospital services used, including clinics and emergency room visits, will be extracted from the hospital administrative systems. | for 12 months

SECONDARY OUTCOMES:
Evaluated health outcomes composite (functional status, symptom intensity) - The functional status will be measured by the Palliative Performance Scale (PPS )(appendix 6). | 12 months
  The PPS is a clinical tool commonly used in the local settings. The level of physical performance is rated on a scale of 100 (normal) to 0 (death), measured in 10 % decrement levels. The scale has been validated and the inter-rater reliability between doctors and nurses maintained at .85 with strong kappa values of .97 (Myers J, Gardiner K, Harris K et al., 2010).

OTHER OUTCOMES:
Perceived outcomes composite (quality of life, caregiver burden, satisfaction with care) | 12 months
  Quality of life will be measured by an ESRF-specific quality of life measure. The caregiver burden will be measured by the Zarit Caregiver Burden Scale (ZCBS). Satisfaction with care will be measured by the 15-item questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth Hospital, Hong Kong, Hong Kong SAR, Hong Kong

IPD SHARING:
Plan to Share IPD: No